CLINICAL TRIAL: NCT04227730
Title: Maternal And Neonatal Screening For Group B Streptococci in Fayoum Governrate: A Follow Up Study
Brief Title: MATERNAL AND NEONATAL SCREENING FOR GROUP B STREPTOCOCCI : A Follow up STUDY
Status: Withdrawn | Type: Observational
Why Stopped: COVID 19 Pandemic disabled team involved
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Sahar MY Elbaradie, associate Professor, Fayoum University Hospital
Other Study IDs: FayoumEgypt
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Group B Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: group A (+ve GBS) 300 pregnant of gestational age 35-37 weeks were screened by a group B streptococcal (GBS) conventional PCR assay. Patients who were followed till delivery without prolonged rupture of membrane were eligible to enter the study and details with regard to labor and delivery were recorded. Infant data were also recorded.
  Interventions: Diagnostic Test: culture and PCR for group B streptococcus
- group B: group B (-ve GBS) 300 pregnant of gestational age 35-37 weeks were screened by a group B streptococcal (GBS) conventional PCR assay. Patients who were followed till delivery without prolonged rupture of membrane were eligible to enter the study and details with regard to labor and delivery were recorded. Infant data were also recorded.
  Interventions: Diagnostic Test: culture and PCR for group B streptococcus

INTERVENTIONS:
Diagnostic Test: culture and PCR for group B streptococcus — all participants were evaluated by vaginorectal specimens for the detection of GBS, The swabs are placed in Amies transport medium and sent to the microbiology laboratory for testing by conventional PCR assay.

SUMMARY:
Group B Streptococcus (GBS), is a facultative gram positive diplococcus originally known for causing bovine mastitis and was not demonstrated to be a human pathogen until 1938. In the 1970s, GBS emerged as the leading cause of neonatal morbidity and mortality, with a frequency of 2-3 cases per 1,000 live births and case-fatality ratios as high as 50%

DETAILED DESCRIPTION:
Group B Streptococcus (GBS), is a facultative gram positive diplococcus originally known for causing bovine mastitis and was not demonstrated to be a human pathogen until 1938 (1). In the 1970s, GBS emerged as the leading cause of neonatal morbidity and mortality, with a frequency of 2-3 cases per 1,000 live births and case-fatality ratios as high as 50% (2). It causes severe invasive infection in newborns 80% of which occur within the first week of life (early-onset neonatal sepsis) that results from ascending spread of GBS into the amniotic fluid through both ruptured and intact membranes (3,4). Infants who have such infections may require prolonged hospitalization, and those who survive may have mental retardation or visual loss (5).

Transmission from mother to child has been reported to be 29 times higher in GBS-colonized mothers than in noncolonized mothers. The prevalence of GBS colonization in the vagina and/or rectum among pregnant women can vary among ethnic groups and geographical locations, ranging from approximately 10% to 40% (6). Although GBS colonization is not associated with disease in healthy women, colonization in pregnant women may be associated with urinary tract infection, bacteremia, amnionitis, endometritis, postpartum wound infections, and rarely, meningitis (7).

A number of obstetric factors have been associated with an increased likelihood of early-onset GBS disease in the newborn. These include maternal colonization of the vagina and rectum with GBS, preterm birth, prolonged rupture of membranes, intrapartum fever, women younger than 20 years (8), women with prior GBS-infected infant, women with heavy colonization- GBS bacteriuria equal to or greater than 104 colony forming units or low levels of anti-GBS capsular antibody(9,10).

Intrapartum antibiotic prophylaxis (IAP) has been shown not only to interrupt the transmission of GBS from mother to infant but also to reduce the incidence of early-onset GBS disease (11). Guidelines from the Federal Centers for Disease Control and Prevention (CDC) (12), the American College of Obstetricians and Gynecologists (ACOG) (6) and the American Academy of Pediatrics (AAP) issued in 1996 and 2002(13, 14) recommended two different strategies for the selection of candidates for IAP: either screening for GBS vaginorectal carriers or identification of maternal clinical risk factors for early-onset neonatal GBS disease. They recommended obtaining rectovaginal cultures at 35-37 weeks of gestation with the culture-based approach (12).

The value and practicality of both strategies has been debated in the literature. At issue is potential overtreatment (in the case of the culture strategy) and under treatment (in the case of the risk-factor strategy) of patients, as well as the associated cost. For example, the standard screening test, a rectovaginal culture taken at 35 to 37 weeks, has been controversial because it may not accurately predict genital tract colonization at time of labor (with an estimated sensitivity of 87%-91% and specificity of 89%-96%). The risk-factor method, on the other hand, would target treatment toward the mothers believed to be at greatest risk but would miss many colonized mothers and at-risk infants (15, 16). Despite their limitations, both approaches are effective in reducing early-onset group B streptococcal infection rate in infants, although more widespread implementation of the guidelines is needed (11, 17).

The Committee on Obstetric Practice 2003 recognized that compliance with the culture-based approach will require the implementation of several steps (18)

* Obtaining accurate culture media
* Appropriate processing of the culture by laboratories
* Timely reporting of results to obstetric providers
* Administering intrapartum prophylaxis to culture-positive women

The sensitivity of cultures in detecting GBS colonization varies from 54% to 87%, and results has a slow turnaround time requiring up to 36 to 72 hours before results can be issued(3,16). Besides being time-consuming, this method requires an experienced technician to identify the suspected colonies, which are not always beta-hemolytic. Moreover, the suppression of GBS growth by enterococci present in the vaginal and rectal flora could lead to false-negative results (19).

Rapid methods of detection of GBS colonization in pregnant women namely molecular biology based assays have become the focus of investigation in recent years. The most promising of these techniques is the polymerase chain reaction (PCR), which is reported to be highly sensitive and specific among women in labor and to yield results in 30 to 45 minutes (20).

The rate of GBS colonization and disease among pregnant women and their infants has not been studied in Egypt, and no preventive strategy has been formulated with regard to intrapartum antimicrobial prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* pregnant females 35-37 weeks of gestational age Patients who were followed till delivery without prolonged rupture of membrane

Exclusion Criteria:

* patients lost follow up and or had prolonged rupture of membrane>12 hours

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant females 35-37 weeks of gestational age attending the antenatal outpatient clinic at AlFayom University Hospital. All participants were screened by a group B streptococcal (GBS) conventional PCR assay. Patients who were followed till delivery without prolonged rupture of membrane were eligible to enter the study and details with regard to labor and delivery were recorded delivery was conducted at AlFayom university hospital. Infant data were also recorded.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
prevalence of GBS in Fayoum | one year
  Percentage of maternal GBS infection and its reflection on neonatal infection

SECONDARY OUTCOMES:
improve and simplify the diagnosis of GBS | one year
  Rapid methods of detection of GBS colonization (molecular biology based assay) the polymerase chain reaction (PCR),

CONTACTS AND LOCATIONS:
Locations (1):
- sahar M.Y elbaradie, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided